CLINICAL TRIAL: NCT00570882
Title: A Randomized Phase II Trial Of Sunitinib Administered Daily For 4 Weeks, Followed By 2-Week Rest Vs. 2-Week On And 1-Week Off In Metastatic Renal Cell Carcinoma
Brief Title: Study of Sunitinib Administered as 4/2 vs. 2/1 Schedule in Advanced Renal Cell Carcinoma (RCC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Responsible Party: Principal Investigator, JLee, Associate professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UOSG_AMC_0701
Record Dates: First submitted 2007-12-10; First posted 2007-12-11 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Metastatic Renal Cell Carcinoma
Keywords: Renal cell carcinoma; Sunitinib; phase II study; Randomized study
MeSH Terms: conditions — Carcinoma, Renal Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sunitinib 4/2 (Active Comparator): Sunitinib 50 mg PO 4-week on and 2-week off
  Interventions: Drug: Sunitinib 4/2
- Sunitinib 2/1 (Experimental): Sunitinib 50 mg PO 2-week on 1-week off
  Interventions: Drug: Sunitinib 2/1

INTERVENTIONS:
Drug: Sunitinib 2/1 — Sunitinib 50 mg PO 2 weeks followed by 1 week rest
  Arms: Sunitinib 2/1
Drug: Sunitinib 4/2 — Sunitinib 50 mg PO 4 weeks followed by 2 week rest
  Arms: Sunitinib 4/2

SUMMARY:
This study is to evaluate the efficacy, safety, and feasibility of sunitinib in 4/2 and 2/1 regimen in previously untreated metastatic RCC to select the most promising regimen, which should be used in further studies of this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically confirmation of renal cell carcinoma with a clear cell histologic component
2. Patients must present with stage IV disease not amenable to surgery, radiotherapy, or combined modality therapy with curative intent.
3. Measurable disease according to RECIST criteria are required but patients with evaluable lesions without measurable lesions are allowed to be enrolled to this study
4. ECOG performance status 2 or better
5. Age 18 years or older
6. Adequate bone marrow, hepatic, and renal function
7. Life expectancy of > 3 months
8. Singed and dated informed consent of document indicating that the patient (or legally acceptable representative) has been informed of all pertinent aspects of the trial prior to enrollment

Exclusion Criteria:

1. Known spinal cord compression or carcinomatous meningitis
2. Diagnosis of any serious secondary malignancy within the last 2 years, except for adequately treated basal cell or squamous cell carcinoma of skin, or in situ carcinoma of cervix uteri
3. Hypertension that cannot be controlled by medications (blood pressure > 150/90 mmHg despite optimal medical therapy)
4. Treatment with anticonvulsant agents and treatment with therapeutic doses of coumadin currently or within 2 weeks prior to first day of sunitinib administration. Low dose coumadin for DVT prophylaxis is permitted (up to 2 mg/day).
5. Pregnancy or breast feeding.
6. Other severe acute or chronic medical or psychiatric condition
7. Prior treatment on sunitinib, sorafenib, or bevacizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2007-10; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Treatment failure rate (progressive disease, treatment withdrawal due to unacceptable toxicities, or any death) | 12 months
  From the date of randomization to the date of progressive disease, treatment withdrawal, or death from any cause, which came first.

SECONDARY OUTCOMES:
Overall response rate | 6 months
  RECIST v.1.1 will be used to assess tumor responses
quality of life | 12 months
  EORTC QLQ C30 and EQ5D will be used to assess the quality of life
Progression free survival | 12 months
Overall survival | 36 months
Adverse events | about 12 months
  CTC AE v.3.0

CONTACTS AND LOCATIONS:
Overall Officials: Jae-Lyun Lee, MD, PhD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Daegu Catholic University Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Asan Medical Center, Seoul

REFERENCES:
- [Derived] Lee JL, Kim MK, Park I, Ahn JH, Lee DH, Ryoo HM, Song C, Hong B, Hong JH, Ahn H. RandomizEd phase II trial of Sunitinib four weeks on and two weeks off versus Two weeks on and One week off in metastatic clear-cell type REnal cell carcinoma: RESTORE trial. Ann Oncol. 2015 Nov;26(11):2300-5. doi: 10.1093/annonc/mdv357. Epub 2015 Sep 7. PMID 26347107